CLINICAL TRIAL: NCT02670200
Title: MAC-CBT Used as Internet-delivered Psycho-oncological Support
Brief Title: Internet-delivered Psycho-oncological Support
Acronym: ICBT_MAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuropsychiatrischen Zentrums Hamburg-Altona (Other)
Collaborators: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Peter Tonn, Managing director of the Department, Neuropsychiatrischen Zentrums Hamburg-Altona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NS-2016-001
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cancer
Keywords: psychooncology; mental health support; ICBT; supportive treatment for cancer patients; depression; online-therapy; Psycho-oncological support via internet; internet-delivered cognitive behavior medicine
MeSH Terms: conditions — Neoplasms; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm / verum arm (Experimental): Participants can work on ten modules specialized cognitive behavior treatments to learn and deal with mindfulness, acceptance and commitment. They should learn to handle their emotions, to accept the situation and to get in an active future. The participants can direct contact a psychotherapist via email, Chat or Skype/tokbox. The modules based on Cognitive Behavior Therapy.
  Interventions: Behavioral: cognitive behavior therapy
- non-intervention arm / control group (Active Comparator): Participants can work on six modules with information und education goals for learning something about their possibilities to become a better mood, better psychovegetative or psychosocial situation as cancer patient. This modules are based on Cognitive Behavior Therapy. The non-intervention arm will only allow contact to the platform, no direct contact to a psychotherapist (in opposite to the intervention arm) is available.
  Interventions: Behavioral: cognitive behavior therapy

INTERVENTIONS:
Behavioral: cognitive behavior therapy — treatment technique to help people to overcome psychological distress and mental diseases

SUMMARY:
Cancer patients develop a high psychological burden of the underlying disease. To support patients in outpatient phases psychotherapists are not sufficiently available for establish regularly face-to-face-contact. The availability of Internet-based psychotherapeutic support can bridge this gap. This study examines the effectiveness of MAC-CBT® via the Internet (called Incobeth®) in cancer patients.

DETAILED DESCRIPTION:
In this study, a randomized trial is conducted in which the online users are allocated into two different care services (MAC-CBT® vs. psycho-educational support program). Participants are cancer patients who have been advised by their treating oncologists, family doctors or psychotherapists on the online support. All patients are randomized, based on the information the referring physician give about type of tumor, treatment status, prognosis and psychosocial factors. Initial will be done an extensive psychometric survey. The MAC-CBT® group receives an intervention program based on ten modules, in which the aspects of Mindfulness, Acceptance and Commitment in detail are included to start a process-oriented self-treatment with regular feedback by the individually assigned psychologists through the internet-portal and email and through live contacts (via video-telephony). The control group will have access to six modules with a psychoeducational support program, which is also constructed according to the MAC principle. Both groups can use crisis modules (in case of pain, psychological crisis, fear of dying) without access restriction. The control group, upon completion of 6 weeks (for each module one week) can switch to active treatment arm. Input and output results are determined using validated survey instruments. Randomisation is done by a physician not involved in the further course of the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patient
* psychological distress
* informed consent

Exclusion Criteria:

* no informed consent
* no cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Scores of Prime-MD | Start at baseline (t1), Second measurement at t2 estimated 8 weeks later, Followup 6months (t3)
  Recording of change of score PRIME-MD, depression, anxiety and other mental health issues

SECONDARY OUTCOMES:
Scores of Quality of Life | Start at baseline (t1), Second measurement at t2 estimated 8 weeks later, Followup 6months (t3)
  Measurement of the changes of quality of life after the treatment
Resilience | Start at baseline (t1), Second measurement at t2 estimated 8 weeks later, Followup 6months (t3)
  Reflection of the changes of resilience to test if it is stable or fluid over the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tonn, MD, Principal Investigator — Managing Director
Locations (1):
- Neuropsychiatric Center of Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
No this ist not planned yet.